CLINICAL TRIAL: NCT01594541
Title: Hyperhomocysteinemia in a Mild Cognitive Impairment and Dementia Population: the Effect of Treatment With Cerefolin NAC® in a Naturalistic Community-based Dementia Practice
Brief Title: A Retrospective Analysis of Cerefolin NAC® in Cognitively Impaired Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pamlab, Inc. (Industry)
Collaborators: Clionsky Neuro Systems Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NAC-004
Record Dates: First submitted 2012-04-03; First posted 2012-05-09 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Mild Cognitive Impairment
Keywords: hyperhomocysteinemia; dementia; depression; vitamin B12; mild cognitive impairment; alzheimer's
MeSH Terms: conditions — Cognitive Dysfunction; Hyperhomocysteinemia; Dementia; Depression

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients Treated with CerefolinNAC®
- Patients Not Treated with CerefolinNAC®

SUMMARY:
This retrospective analysis of de-identified data from 700 charts of consecutive patients from this patient population is to investigate the prevalence of hyperhomocysteinemia and associated metabolic abnormalities in this naturalistic grouping of patients with various stages of cognitive loss and diagnosed with various types of dementia.

DETAILED DESCRIPTION:
A single-center, retrospective review of the medical charts of 700 de-identified elderly patients who underwent evaluation and treatment for cognitive loss including analysis of:

Laboratory values of interest: homocysteine, methylmalonic acid, CRP, BNP, CO2, TSH, Fe/TIBC, RPR/TPPA/FTA-ABS, and if available, folic acid and B12 levels ordered by primary care providers.

Neuropsychological tests of executive function, memory and affect:

* Wechsler Memory Scale-Revised (WMS-R) or Fourth Edition (WMS-IV)

  * Logical Memory -Delayed Recall, Scaled Score
  * Visual Reproduction-Delayed Recall, Scaled Score
* Shopping List Test, Delayed Recall
* Trailmaking A and B Tests
* Verbal Absurdities subtest of the Stanford Binet, Form L-M
* Proverbs Test
* Memory Orientation Screening Test
* Folstein Mini-Mental State Exam
* Geriatric Depression Scale, 15 items

Sub-group analysis of MRI volumetrics and PET scans when available. Sequentially pulled from June 1, 2009 to September 2011

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 55 and 89 years old
* Meeting criteria for Mild Cognitive Impairment or dementia with a minimum MOST score of 5 but not over 23
* Has a minimum of 3 months evaluation
* Able to undergo testing for cognition and complete the GDS

Exclusion Criteria:

* Known allergy/intolerance to any ingredient in Cerefolin NAC®
* Substantial impediments to adherence, such as severe dementia without caregiver to administer medication
* Inability to swallow pill-form medication
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease
* Hcy score lower than 11

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical charts of 700 de-identified elderly patients who underwent evaluation and treatment for cognitive loss.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Levels of Homocysteine Over Time | Week 6, Week 12, and Quaterly Thereafter @ 6 Month Intervals
  To analyze homocysteine levels, cognitive test scores and depression level to determine the prevalence of hyperhomocysteinemia and associated metabolic abnormalities and compare results of patients on Cerefolin NAC® alone to patients on Cerefolin NAC® in combination with standard of care memory and/or depression medications.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of Cerefolin NAC® based on adverse events, discontinuation due to intolerability and compliance. | Baseline, Week 6, Week 12, and Quarterly Thereafter @ 6 Month Intervals
Examine the demographics, medical co-morbidities present and affective and cognitive characteristics of the group of patients demonstrating hyperhomocysteinemia compared with the group without hyperhomocysteinemia in a dementia population. | Baseline, Week 6, Week 12, and Quarterly Thereafter @ 6 Month Intervals

CONTACTS AND LOCATIONS:
Overall Officials: Emily Clionsky, MD, Principal Investigator — Clionsky Neuro Systems Inc.
Locations (1):
- Clionsky Neuro Systems, Inc., Springfield, Massachusetts, United States